CLINICAL TRIAL: NCT00396162
Title: Use of Probiotics as Adjunctive Treatment for Chronic Rhinosinusitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Institut Rosell (Other)
Responsible Party: Principal Investigator, Jeffrey E. Terrell, M.D., Professor of Otolaryngology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00006212
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Results first posted 2016-08-04 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Rhinosinusitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo pill (Placebo Comparator): Placebo pills on same schedule as active intervention.
  Interventions: Other: Placebo
- Probiotic (Active Comparator): L. rhamnosus R0011 strain
  Interventions: Drug: probiotic containing L.rhamnosus R0011 strain

INTERVENTIONS:
Drug: probiotic containing L.rhamnosus R0011 strain — 500 million active cells of L rhamnosus R0011 strain per tablet bid for 4 weeks
  Other Names: L rhamnosus R0011
  Arms: Probiotic
Other: Placebo — Placebo pill
  Arms: Placebo pill

SUMMARY:
Chronic sinusitis is reported to be one of the most widespread disorders in the United States. It can be caused by a variety of reasons such as allergy, infection and/or defects in T-cells which help regulate immune function. Medication and other costs related to treatment of nasal and sinus infections are estimated to be more than $60 million annually putting a considerable strain on the economy of health care.

Probiotics are live microorganisms that are normally present in the gut of a healthy individual. They are also known as "friendly bacteria" and have been used to help maintain the normal functioning of the immune system. They are safe and are commercially available in the form of yoghurt, sachets, chewable tablets or flavored capsules. Since a number of nasal and sinus disorders are related to allergy and improper functioning of the immune system, we hypothesize that regular use of probiotics may help improve chronic nasal and sinus symptoms by boosting immune responses.

The project we propose is novel because it would be the first study evaluating the usefulness of probiotics for the larger population having chronic sinusitis rather than those having only allergic symptoms. We aim to assess whether regular use of probiotics will help improve symptoms of chronic sinusitis and will have a greater effect than placebo in this regard.

DETAILED DESCRIPTION:
Probiotics are live microorganisms which when administered in adequate amounts confer a health benefit on the host. They are a part of the normal gastrointestinal flora and have safely been used to boost immune responses in patients with perennial and seasonal allergic rhinitis. Their exact mechanism of benefit is unknown but they primarily help to regulate T-cell function which is important in maintaining immune tolerance.

Chronic rhinosinusitis is widely prevalent and affects nearly 16 million people in the US alone each year. It puts a strain on the health resources of the nation in terms of costs related to medications and surgery. Chronic rhinosinusitis can be caused by a variety of reasons including allergy/hypersensitivity, infection, nasal anatomical variations and T-cell regulatory dysfunction. We hypothesize that regular use of probiotics in patients with chronic rhinosinusitis will result in substantial improvement in their symptoms by boosting their immunity and may also help decrease their medication usage.

Our study will be a double-blinded, randomized, control trial. We hope to recruit 100 patients from the University Otolaryngology and Allergy Clinics. Fifty patients will be randomized to the treatment (active) arm and 50 patients to the placebo arm. Subjects will be followed for 2 months during their period of participation in the study.

The main aim of our study is to determine whether regular use of probiotics in patients with chronic rhinosinusitis helps improve their quality of life. Our main outcome of interest is a change in the mean score of the Sino-Nasal Outcome Test (SNOT-20) form in the treatment group and a greater change in the mean score of the SNOT-20 in the treatment arm as compared to the placebo arm. If probiotics are found to be effective, they may be used as a cost-effective, adjunctive therapy for patients with chronic rhinosinusitis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥15 and ≤70 years.
2. The patient must be bothered by each of the two following symptoms(>50% of days in the last 3 months):

   A. More than 12 consecutive weeks of symptomatic nasal obstruction and, B. More than 12 weeks of symptomatic nasal discharge.
3. An Otolaryngologist evaluation and diagnosis of chronic inflammatory rhinosinusitis (hyperplastic mucosa, polyps in absence of overt bacterial infection)
4. Access to telephone (home or person cell).

Exclusion Criteria:

1. Sinus surgery within the last 3 months
2. Acute illness within the last 2 weeks requiring antibiotics: including: otitis media, pharyngitis, bronchitis, or laryngitis.
3. Immunosuppression (due to medications including oral steroids, or due to autoimmune diseases, HIV infection, cystic fibrosis, immunodeficiency, malignancies, uncontrolled diabetes mellitus, chronic renal failure, etc.)
4. Patients with chronic or acute bacterial sinusitis.(Clinical diagnosis-to be decided by MD)
5. An allergic reaction to a probiotic dietary supplement in the past (such as symptoms of tightness in the chest, breathing difficulties, skin hives, rash or other clinical symptoms consistent with sensitivity or intolerance)
6. Inability to speak or read English.
7. Pregnancy and Lactation

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2006-11; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey E Terrell, MD, Principal Investigator — University of Michigan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 82 participants were screened . 77 enrolled.
Groups:
- Probiotic: The study protocol scheduled daily oral supplementation of either the probiotic or the placebo twice daily for four weeks. The probiotic product was a chewable tablet containing 500 million active cells of L rhamnosus R0011 strain per tablet. Placebo tablets comparable to the probiotic in color, weight, texture, and flavor were also available.
- Placebo: Placebo tablets comparable to the probiotic in color, weight, texture, and flavor were also available.
Period: Overall Study
Arm/Group | Probiotic | Placebo
Started | 39 | 38
Completed | 37 | 35
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Probiotic: drug
  probiotic containing L.rhamnosus R0011 strain: 500 million active cells of L rhamnosus R0011 strain per tablet bid for 4 weeks
- Placebo Pill: Placebo pills on same schedule as active intervention.
  probiotic containing L.rhamnosus R0011 strain: 500 million active cells of L rhamnosus R0011 strain per tablet bid for 4 weeks
- Total: Total of all reporting groups
Arm/Group | Probiotic | Placebo Pill | Total
Number analyzed (Participants) | 39 | 38 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (12.6) | 49.6 (8.6) | 49.5 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 25 | 44
  Male | 20 | 13 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 37 | 35 | 72
  Unknown or Not Reported | 0 | 0 | 0
asthma [Number; unit: participants]
  No asthma | 14 | 14 | 28
  intermittent and mild asthma | 13 | 10 | 23
  moderate-severe asthma | 12 | 14 | 26
aspirin sensitivity [Number; unit: participants]
  Aspirin Sensitivity | 12 | 12 | 24
  No aspirin sensitivity | 27 | 26 | 53
SinoNasal Outcome Test Score (SNOT-20) [Mean (Standard Deviation); unit: units on a scale] — SinoNasal Outcome Test measures symptom severity. It is a summary score, ranging from 0 to 100 with 100 indicating worse symptoms.
  units on a scale | 36.4 (16.2) | 39.5 (19.8) | 37.9 (17.9)

OUTCOME MEASURES:

1. Primary Outcome: Mean Reduction in SNOT-20 Scores
Description: Mean reduction (and Standard deviation) in SNOT-20 scores, from baseline to 8 week measurements. SinoNasal Outcome Test measures symptom severity. It is a summary score, ranging from 0 to 100 with 100 indicating worse symptoms. Since 100 represents more severe symptoms, the changes represented here are reductions in SNOT-scores, even though they are not expressed as negative numbers.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Probiotic | Placebo
Number analyzed (Participants) | 37 | 35
units on a scale | 1.8 (12) | 5.5 (14)
Statistical Analysis 1: Comparison: Probiotic vs Placebo; Test type: Superiority or Other; p = 0.23, t-test, 2 sided

2. Secondary Outcome: Side Effect Summary
Description: Totals of all side effects for placebo group and treatment group over the course of the eight week trial (including patients who dropped from the study after baseline measurement). Individual categories of side-effects are listed in Adverse events section.
Time Frame: 8 weeks
Population: The sample size on the placebo side is reduced due to some study participants not reporting their 8 week survey
Measure: Number; unit: participants
Arm/Group | Placebo Pill | Probiotic
Number analyzed (Participants) | 35 | 37
participants | 17 | 14
Statistical Analysis 1: Comparison: Placebo Pill vs Probiotic; Test type: Superiority or Other; p = .31, t-test, 2 sided

3. Secondary Outcome: Mean Number of Days of Antibiotic Use During the Study Period (0-8 Weeks)
Description: Mean number of days that antibiotics were used in the subgroup (placebo vs Probiotic arm)
Time Frame: At 8 weeks after baseline measures
Measure: Mean (Standard Deviation); unit: days
Groups:
- Active Intervention: The study protocol scheduled daily oral supplementation of either the probiotic or the placebo twice daily for four weeks. The probiotic product was a chewable tablet containing 500 million active cells of L rhamnosus R0011 strain per tablet. Placebo tablets comparable to the probiotic in color, weight, texture, and flavor were also available.
Arm/Group | Placebo | Active Intervention
Number analyzed (Participants) | 35 | 37
days | 1.9 (5.5) | 0.8 (2.7)

4. Secondary Outcome: Mean Number of Days of Steroid Spray Use for Each Group
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Probiotic | Placebo
Number analyzed (Participants) | 37 | 35
days | 2.8 (7.4) | 0.4 (2.2)

ADVERSE EVENTS:
Arm/Group | Active Intervention | Placebo
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/38
Other Adverse Events (participants affected / at risk) | 14/39 | 17/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Intervention (N=39) | Placebo (N=38)
bloating (Gastrointestinal disorders) | 7 | 9
diarrhea (Gastrointestinal disorders) | 8 | 10
abdominal pain (Gastrointestinal disorders) | 7 | 7
loose stools (Gastrointestinal disorders) | 9 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No